CLINICAL TRIAL: NCT05211089
Title: Comparison of Manual Versus Automated Choroidal Thickness Measurements Using Swept-source Anterior Segment Optical Coherence Tomography
Brief Title: Manual Versus Automated Choroidal Thickness Measurements Using Swept-source Anterior Segment OCT
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate professor of Ophthalmology, Assiut University
Other Study IDs: 17300719
Record Dates: First submitted 2022-01-25; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Eye Diseases
Keywords: Choroidal thickness; Swept source; OCT
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Optical Coherence Tomography imaging of choroid — A single expert retinal specialists used a Topcon DRI-1 SS-OCT to do the Choroidal Thickness measurements. A 12, 9-mm radial line scan procedure was performed. Each radial line was automatically scanned 32 times in the same spot, followed by the creation of 12 high-resolution average B-scan images. Each scan was double-checked to confirm that it was centred on the fovea. Only scans of good quality were included. The perpendicular distance between the outer border of the RPE and the junction of the choroid and sclera was used to calculate CT. It was calculated automatically using the mapping software incorporated into the device and displayed as a colourful topographic map with nine subfields defined by the Early Treatment Diabetic Retinopathy Study (ETDRS) style grid.

SUMMARY:
The choroid, which is located between the retina and the sclera, is a connective tissue layer that is densely packed with blood vessels and is responsible for supplying oxygen and nutrients to the retina's periphery. One of the primary functions of the choroid is to support the metabolism of the retinal pigment epithelium (RPE). It is implicated in the pathogenesis of a variety of retinal disorders, including age-related macular degeneration, polypoidal choroidal vasculopathy, central serous chorioretinopathy, and high myopia-associated chorio retinal atrophies. Because choroidal alteration has a fundamental role in the development and progression of these diseases, choroidal thickness provides comprehensive information to physicians.

For the study of the choroid, researchers have used ultrasound, magnetic resonance imaging MRI, and Doppler laser, but these methods have limited utility due to a lack of resolution. Contrary to this, indocyanine green (ICG) angiography provides valuable clinical information but does not provide cross-sectional images of the choroid for in vivo research studies.

Optical coherence tomography (OCT) has gained in popularity in clinical and experimental ophthalmology over the last decade as a way to acquire detailed, three-dimensional images of the retina . Imaging the entire choroid, on the other hand, has proven to be more difficult due to the significant decline in signal strength beyond the RPE prompted by the pigment in the RPE and choroid and light scattering in the vasculature. The development of improved depth imaging (EDI) by Spaide et al. opened the door to quantitative choroid assessment. Choroid imaging is currently possible using one of two optical coherence tomography (OCT) techniques: (1) spectral-domain (SD) OCT utilizing standard light sources using EDI, and (2) swept-source (SS) OCT using a long wavelength light .A 1 m-band light source is used in SS-OCT, which penetrates deeper into the retino choroidal tissues and so optimizes the resolution. To better visualize retinal and choroidal changes, SS-OCT can concurrently display a focused image of both the retina and the choroid. This renders it an accurate technology for assessing choroidal thickness.

Such findings of choroidal thickness changes revealed that the choroid and choroidal thickness may be important attributes in the evaluation of ocular pathology. To properly understand the scientific value of these potential choroidal thickness variations, it would appear that comprehensive and systematic normative values for choroidal thickness are fundamental.

ELIGIBILITY:
Inclusion Criteria:

* Normal adult volunteers

Exclusion Criteria:

* Eyes with chorioretinal or vitreoretinal diseases
* History of intraocular surgery
* Glaucoma.
* Systemic diseases or conditions that could affect retinal or choroidal thickness,
* Pregnant women

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Normal adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Choroidal thickness | 1 day
  Manual and automated measurement of choroidal thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No